CLINICAL TRIAL: NCT01171196
Title: Validation of Questionnaires to Identify Chinese Patients at Risk for Obstructive Sleep Apnea
Brief Title: Questionnaires to Identify Chinese Patients at Risk for Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Agnes Yuen-Kwan Lai, Senior Technical Officer, The University of Hong Kong
Other Study IDs: HKCTC-1117
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Last update posted 2015-11-09 (Estimated); Status verified 2015-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Sleep Apnea; Questionnaire
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to validate the Berlin questionnaire and STOP-BANG (snore, tired, obstruction, pressure, body mass index (BMI), age, neck, gender) as effective screening tools for Chinese subjects who are suspected to have obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common sleep related breathing disorder associated with excessive daytime sleepiness and cardiovascular disease. It is prevalent in both western (4-26%) and eastern countries (4-19%). In recent studies, it has been estimated that at least 70-80% of middle aged individuals with sleep apnea are undiagnosed and untreated. The prevalence of undiagnosed OSA subjects within the community suggests the need for a greater awareness and a high index of suspicion of this disease entity as well as its associated short- and long-term comorbidities.

A reliable and easy-to-use screening questionnaire is required for efficient prediction of OSA and treatment arrangement. It would be helpful to prioritize patients who require sleep study according to the probability of suffering from sleep apnea. It reduces the use of sleep study for those with low probability of having OSA, but giving treatment to those who are with more severe OSA first. Meanwhile, it enhances the cost effective management of disease especially with limited resources in our society.

ELIGIBILITY:
Inclusion Criteria:

a. No known history of any sleep disorder

Exclusion Criteria:

1. History of heavy alcoholism ( ≥ 3 times / week)
2. Underlying pulmonary diseases
3. Recent upper respiratory tract infection in the past one week
4. Unstable medical conditions
5. Pregnancy
6. History of psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who are referred to have a diagnostic polysomnography (PSG) will be recruited from the Sleep Disorders Centre, Department of Medicine, Queen Mary Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2010-07; Primary Completion 2014-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
To validate the Berlin questionnaire and STOP-BANG as effective screening tools | at the time of completing the questionnaire
  To validate the Berlin questionnaire and STOP-BANG as effective screening tools for Chinese subjects who are suspected to have OSA

SECONDARY OUTCOMES:
the predictive performance on OSA of Berlin questionnaire and STOP-BANG | at the time of completing questionnaire
  To compare the predictive performance on OSA of Berlin questionnaire and STOP-BANG in our Chinese population

CONTACTS AND LOCATIONS:
Overall Officials: Agnes YK Lai, MSc, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong Island, Hong Kong, Hong Kong